CLINICAL TRIAL: NCT02157493
Title: Evaluation of an Entrepreneurship Program on Psychosocial, Behavioral Health, Educational and Economic Outcomes Among American-Indian Youth
Brief Title: Evaluation of an Entrepreneurship Program for American-Indian Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Native American Research Center for Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: U261IHS0080-01-00
Record Dates: First submitted 2014-06-04; First posted 2014-06-06 (Estimated); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Depressive Symptoms; Substance Use
Keywords: American Indian; Adolescents; Entrepreneurship; Paraprofessional; Life skills
MeSH Terms: conditions — Depression; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arrowhead Business Group Curriculum (Experimental): The Arrowhead Business Group (ABG) Curriculum is a 22-session youth entrepreneurship/life-skills intervention delivered by trained American Indian paraprofessionals from the community to mixed-gender groups of approximately 25 youth. The intervention is delivered over a 3 night/4 day camp along with weekend workshops once a month for 6 months during the academic year. Depending on the time of enrollment, subjects will receive follow-up assessments at 6-month intervals for up to 36-months post-intervention. (Subjects in this cohort will also receive the activities associated with the control condition.)
  Interventions: Behavioral: Arrowhead Business Group Curriculum; Behavioral: Recreational League Control Condition
- Recreational League Control Condition (Active Comparator): The Recreational League Control Condition will be led by local American Indian study staff who are experienced with Johns Hopkins camps and community-based Apache sports programs. Sports and recreational activities will be conducted on 3 Saturdays during the academic year to mixed gender groups of approximately 50 participants.
  Interventions: Behavioral: Recreational League Control Condition

INTERVENTIONS:
Behavioral: Arrowhead Business Group Curriculum — Arrowhead Business Group (ABG) is a culturally tailored entrepreneurship/life-skills intervention, which features instruction from American Indian paraprofessionals in an effort to decrease drug use, depressive symptoms, hopelessness and other high-risk behaviors among youth while improving their school performance and college/career aspirations.
  Arms: Arrowhead Business Group Curriculum
Behavioral: Recreational League Control Condition — The control condition will consist of a recreational sports league that will be led by local American Indian study staff who are experienced with Johns Hopkins camps and community-based Apache sports programs. Activities will be conducted on 3 Saturdays during the academic year to mixed gender groups of approximately 50 participants.

SUMMARY:
This study will use a randomized controlled design to evaluate whether a youth entrepreneurship/life-skills intervention for reservation-based American Indian adolescents (ages 13-15) improves psychosocial, behavioral health, educational, and economic outcomes from baseline for up to 3 years follow-up as compared to a recreational sports league control condition.

DETAILED DESCRIPTION:
Intervention activities will be held over a 3 night/4 day residential camp and 6 weekend workshops during the academic year. The control condition will consist of a recreational sports league held on 3 Saturdays, also during the academic year.

ELIGIBILITY:
Inclusion Criteria:

* American Indian ethnicity and primary residence within the Fort Apache Indian Reservation.
* Participants must be 13-15 years old, enrolled as a student at one of the participating high schools, and must have parent/guardian consent for participation in the study.

Exclusion Criteria:

* Youth that are currently enrolled in foster care will not be eligible to participate in the study.
* Those unable to participate in any of the evaluation assessments or intervention components will also be excluded.

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 449 (Actual)
Dates: Start 2014-04; Primary Completion 2018-07 (Actual); Study Completion 2019-06-25 (Actual)

PRIMARY OUTCOMES:
Decreased substance use as measured by Youth Risk Behavior Survey (YRBS) in treatment vs. control group at 24 months follow-up | 24 months follow-up

SECONDARY OUTCOMES:
Decreased depressive symptoms on Patient Health Questionnaire-9 (PHQ-9) in treatment vs. control group at 24 months follow-up | 24 months follow-up
Increased academic achievement as measured by school records and Across Time Orientation measure in treatment vs. control group at 24 months follow-up | 24 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Allison Barlow, PhD, MPH, MA, Principal Investigator — Johns Hopkins Center for American Indian Health
Locations (1):
- Johns Hopkins Center for American Indian Health - Whiteriver Office, Whiteriver, Arizona, United States